CLINICAL TRIAL: NCT01793727
Title: Learning Curve of the Infant Glidescope® Cobalt Video Laryngoscope in Anesthesiology Residents
Brief Title: Infant Glidescope® Learning Curve
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Cengiz Karsli, Primary Investigator, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1000023363
Record Dates: First submitted 2013-02-12; First posted 2013-02-15 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Tracheal Intubation
Keywords: infants; general anesthesia; tracheal intubation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Glidescope intubation (Experimental): Comparison of direct laryngoscopy and Glidescope videolaryngoscopy
  Interventions: Device: Glidescope videolaryngoscope

INTERVENTIONS:
Device: Glidescope videolaryngoscope

SUMMARY:
A prospective trial evaluating the learning curve associated with the use of a videolaryngoscope compared to conventional direct laryngoscopy in infants intubated by anesthesiology residents. Hypothesis: The learning curves of both instruments are equivalent.

ELIGIBILITY:
Inclusion Criteria:

* infants under 10 kg undergoing general anesthesia and requiring tracheal intubation

Exclusion Criteria:

* Difficult airway, severe cardiorespiratory disease, emergency surgery

Max Age: 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2011-07; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Time to optimum visualization of the vocal cords | Under 2 minutes

SECONDARY OUTCOMES:
Time to tracheal intubation | Under 2 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Cengiz Karsli, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada